CLINICAL TRIAL: NCT04780074
Title: Comparative Single-dose Bioavailability Study of Different CoQ10 Formulations in Healthy Adults
Brief Title: Comparative Single-dose Bioavailability Study of Different CoQ10 Formulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Nutrition, Slovenia (Nutris) (Other)
Collaborators: Vizera d.o.o. (Industry); ADM, Ambulanta družinske medicine, Ljubljana, Slovenia (Unknown); Adrialab d.o.o., Ljubljana, Slovenia (Unknown); Tishcon Corp., USA (Unknown)
Responsible Party: Principal Investigator, Igor Pravst, Prof. Dr. Igor Pravst, Institute of Nutrition, Slovenia (Nutris)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TISHCON/CoQ10-01
Record Dates: First submitted 2021-02-23; First posted 2021-03-03 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Bioavailability of Coenzyme Q10
Keywords: coenzyme q10; single dose bioavailability
MeSH Terms: interventions — Methods; I-kappa B Kinase

STUDY DESIGN:
Intervention Model Description: Five-period crossover bioavailability study will include 30 subjects who will test five CoQ10 formulations. Subjects will test 5 formulations of single dose CoQ10 with 2 week wash-out. to assess bioavailability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Standard product (SP): USP CoQ10 powder, hard capsules (Active Comparator): 100 mg per capsule; dosage: 2 capsules - 200 mg total CoQ10
  Interventions: Dietary Supplement: Single dose intervention with Standard product (SP)
- Investigational product 1 (IP1): CoQ10 in soybean oil, softgels (Experimental): 100 mg per softgel; dosage: 2 softgels - 200 mg total CoQ10
  Interventions: Dietary Supplement: Single dose intervention with Investigational product (IP1)
- Investigational product 2 (IP2): Q-Gel hydrosoluble/bioenhanced CoQ10, softgels (Experimental): 100 mg per softgel; dosage: 2 softgels - 200 mg total CoQ10
  Interventions: Dietary Supplement: Single dose intervention with Investigational product (IP2)
- Investigational product 3 (IP3): Qunol Mega Ubiquinol, softgels (Experimental): 100 mg per softgel; dosage: 2 softgels - 200 mg total CoQ10
  Interventions: Dietary Supplement: Single dose intervention with Investigational product (IP3)
- Investigational product 4 (IP4): HydroQsorb Coenzyme Q10, hard capsules (Experimental): 100 mg per capsule; dosage: 2 capsules - 200 mg total CoQ10
  Interventions: Dietary Supplement: Single dose intervention with Investigational product (IP4)

INTERVENTIONS:
Dietary Supplement: Single dose intervention with Standard product (SP) — 2 capsules - 200 mg total CoQ10
  Arms: Standard product (SP): USP CoQ10 powder, hard capsules
Dietary Supplement: Single dose intervention with Investigational product (IP1) — 2 softgels - 200 mg total CoQ10
  Arms: Investigational product 1 (IP1): CoQ10 in soybean oil, softgels
Dietary Supplement: Single dose intervention with Investigational product (IP2) — 2 softgels - 200 mg total CoQ10
  Arms: Investigational product 2 (IP2): Q-Gel hydrosoluble/bioenhanced CoQ10, softgels
Dietary Supplement: Single dose intervention with Investigational product (IP3) — 2 softgels - 200 mg total CoQ10
  Arms: Investigational product 3 (IP3): Qunol Mega Ubiquinol, softgels
Dietary Supplement: Single dose intervention with Investigational product (IP4) — 2 capsules - 200 mg total CoQ10
  Arms: Investigational product 4 (IP4): HydroQsorb Coenzyme Q10, hard capsules

SUMMARY:
The single-center, randomized, open-label, five-period crossover single-dose bioavailability study with five CoQ10 formulations

DETAILED DESCRIPTION:
The single-center, randomized, open-label, five-period crossover bioavailability study will include 30 subjects who will test five CoQ10 formulations. Study will be conducted with single dose CoQ10 to assess bioavailability.

ELIGIBILITY:
Inclusion Criteria:

* Subject Informed consent form (ICF) is singed
* Aged between 18 and 65 years at the time of the signature of ICF
* A body mass index between 18.5-29.9 kg/m2
* Total blood cholesterol range 3,11 - 6,50 mmol/L (not treated with medications)
* Healthy, meaning absence of any prescribed medication for a month prior to the inclusion to the study and during the study
* Willing to avoid a consumption of any food supplements except vitamin D and calcium at least 2 weeks before and during the study
* Consumption of dairy and cereal products (standardised breakfast will include low lactose dairy and bread)
* Willing to follow all study procedures, including attending all site visits (including sessions during which a venous line will be inserted for blood sampling)

Exclusion criteria:

* Intake of any prescribed medication within 2 weeks of the beginning of the study
* Intake of any food supplements within 2 weeks of the beginning of the study, except vitamin D and calcium
* Pregnancy or planned pregnancy
* Breast-feeding mother
* Hypotension
* Any clinically significant history of serious digestive tract, liver, kidney, cardiovascular or haematological disease, diabetes
* Gastrointestinal disorders or other serious acute or chronic diseases
* Known lactose/gluten intolerances/ food allergies (limitation for standardisation of meals)
* Inadequate veins (in the opinion of the investigator) or known contraindication to placement of a dedicated peripheral line for venous blood withdrawal
* Known drug and/or alcohol abuse
* Using any form of nicotine or tobacco
* Mental incapacity that precludes adequate understanding or cooperation
* Participation in another investigational study or blood donation within 3 months prior to or during this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Relative single dose bioavailability (AUC48) of IP (in comparison to SP) | 72 hours
  Relative bioavailability between the investigational products and the standard product (IP1 vs. SP, IP2 vs. SP, IP3 vs. SP, and IP4 vs. SP) expressed as ratio of baseline corrected AUC0-72h, i.e. area under the plasma concentration curve from the administration time to the last observation point (72h) of CoQ10 plasma concentrations above the baseline value.

SECONDARY OUTCOMES:
Relative single dose bioavailability (AUCinf) of IP (in comparison to SP) | 72 hours
  Relative bioavailability between the investigational products and the standard product (IP1 vs. SP, IP2 vs. SP, IP3 vs. SP, and IP4 vs. SP) expressed as ratio of baseline corrected AUCinf, i.e. extrapolated area under the CoQ10 plasma concentration curve above the baseline CoQ10 concentration.

OTHER OUTCOMES:
Relative single dose bioavailability (AUC48) among all the investigational products | 72 hours
  Relative bioavailability among all the investigational products (IP1 vs. IP2, IP1 vs. IP3, IP1 vs. IP4, IP2 vs. IP3, IP2 vs. IP4, and IP3 vs. IP4) expressed as ratio of baseline corrected AUC0-72h, i.e. area under the plasma concentration curve from the administration time to the last observation point (72h) of CoQ10 plasma concentrations above the baseline value.
Relative single dose bioavailability (AUCinf) among all investigational products | 72 hours
  Relative bioavailability among all investigational products (IP1 vs. IP2, IP1 vs. IP3, IP1 vs. IP4, IP2 vs. IP3, IP2 vs. IP4, and IP3 vs. IP4) expressed as ratio of baseline corrected AUCinf, i.e. extrapolated area under the CoQ10 plasma concentration curve above the baseline CoQ10 concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Pravst, Principal Investigator — Nutrition Institute, Ljubljana; Tina Modrej Zadnikar, Principal Investigator — ADM, Ambulanta družinske medicine, Ljubljana, Slovenia
Locations (1):
- ADM, ambulanta družinske medicine, Ljubljana, Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No